CLINICAL TRIAL: NCT00165893
Title: Comparison of Internal Disc Decompression (IDD) vs. a Standardized Non-surgical Treatment Program for Chronic Low Back Pain Secondary to Mild to Moderate Degenerative Disc Disease (DDD)
Brief Title: Comparison of IDD Therapy and Non-surgical Treatment for Low Back Pain Caused by Degenerative Disc Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: North American Medical Corporation (Industry)
Responsible Party: Principal Investigator, Kyle Webb, Research Administrator, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0079-2004
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Degenerative Disc Disease
Keywords: low back pain; DDD
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Physical Therapy Modalities

INTERVENTIONS:
Device: Accu-Spina Device/IDD therapy
Procedure: Physical Therapy

SUMMARY:
This study is looking at a new machine called the Accu-Spina which administers internal disc decompression by following a computer program. This non-surgical treatment (similar to traction) is being compared to a rigorous physical therapy program.

DETAILED DESCRIPTION:
This study is a randomized trial where out of every 3 people, 2 will receive IDD therapy and 1 will have standardized physical therapy. Patients are given surveys to complete that ask about how their back pain is affecting their quality of life before starting treatment, 6 weeks after starting treatment, and 3, 6, and 12 months after starting treatment. If at the 6 week point, the patient and doctor do not think the current treatment is working well enough, the patient is given the option to try the other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain for > 3 months due to mild to moderate disc degeneration, lumbar spondylosis, and facet arthropathy without leg pain based on the physician's history and physical and imaging studies
* Over 18 years old
* Able to provide written informed consent

Exclusion Criteria:

* Infection, neurological deficits, systemic disease that would affect treatment outcome such as inflammatory joint diseases; malignancies with involvement in the musculoskeletal system
* Evidence of severe neural compression on imaging studies, i.e. spinal stenosis or large herniated disc
* Uncontrolled mood disorder
* History of drug or substance abuse
* Lumbar spine pathology requiring surgical intervention
* Previous spine surgery of the lumbar spine, except discectomies >12 months
* Improvement with similar non-surgical treatments in the last 3 months
* Active litigation, workers compensation
* Females whom are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Compare the changes in functional and pain scores in patients with chronic low back pain, which are alternatively treated with a standardized non-surgical treatment program.

SECONDARY OUTCOMES:
Monitoring the side effects, medication use, total charges for treatment, need for continued care, work status, and patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Schaufele, M.D., Principal Investigator — Emory University

REFERENCES:
- See also: Manufacturer's web site with helpful information on IDD therapy. — http://www.iddtherapy.com